CLINICAL TRIAL: NCT04496167
Title: A Phase 2, Randomized, Double Blind, Placebo Controlled Study of the Safety and Efficacy of EN3835 for the Treatment of Adhesive Capsulitis of the Shoulder
Brief Title: Safety and Efficacy of EN3835 in Participants With Frozen Shoulder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EN3835-210
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Adhesive Capsulitis; Frozen Shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EN3835 (Experimental): EN3835 up to 1.74 mg
  Interventions: Drug: EN3835
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EN3835 — Collagenase clostridium histolyticum
  Arms: EN3835
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and efficacy of EN3835 for the treatment of adhesive capsulitis of the shoulder (frozen shoulder).

ELIGIBILITY:
Inclusion Criteria:

1. Have idiopathic unilateral adhesive capsulitis (also known as frozen shoulder).
2. Have unaffected range of motion in the contralateral shoulder as determined by the investigator.
3. Be willing to undergo x-ray and magnetic resonance imaging (MRI) of both affected and unaffected shoulder.
4. Agree to participate in supervised, in-office physical therapy sessions and to complete home exercises at designated time points during the study.
5. Agree to avoid general lifting and carrying during the study as instructed.
6. Be able to read, understand, and independently complete participant reported outcome instruments in English.
7. If female, be of non-childbearing potential (history of hysterectomy, bilateraloophorectomy, bilateral tubal ligation, or postmenopausal with no history of menstrual flow in the 12 months prior to the Screening Visit); or, if of childbearing potential, be non-pregnant, non-lactating and agree to use effective contraception when with a male partner for the duration of the study (and for 28 days after any active treatment period for participant who early terminate). Acceptable forms of contraception include hormonal measures (oral contraceptive pills, contraceptive patch, contraceptive ring, and injections), intrauterine devices, double barrier method (condom plus diaphragm, condom or diaphragm plus spermicidal gel or foam), surgical sterilization of the male partner, and abstinence.
8. If male with reproductive potential, agree to use effective contraception (abstinence, surgical sterilization [vasectomy], or condom with spermicide) with a female partner of child-bearing potential for the duration of the study (and for 28 days after any active treatment period for participant who early terminate).
9. Be willing and able to cooperate with the requirements of the study.
10. Be adequately informed and understand the nature and risks of the study and be able to provide consent .

Exclusion Criteria:

1. Has a known allergy to collagenase or any other excipient of EN3835 or any other procedural medication (including local anesthetics).
2. Has received treatment for adhesive capsulitis (in the timeframes outlined below) or is planning to receive any treatment (other than study treatment) for adhesive capsulitis at any time during the study in the affected shoulder, including but not limited to:

   * Physical therapy or acupuncture within 2 weeks before the first injection of study treatment.
   * Intra-articular or intrabursal injection(s) of lidocaine, suprascapular nerve blocks, or electroanalgesic and/or thermoanalgesic modalities within 1 month before the Screening Visit.
   * Intra-articular or intrabursal injection(s) of corticosteroids within 8 weeks before the Screening Visit.
   * Intra-articular or intrabursal injection(s) of sodium hyaluronate and/or glenohumeral distension arthrography within 3 months before the Screening Visit.
   * Manipulation under anaesthesia at any time prior to the study.
   * Surgery (including arthroscopic or open capsular release, capsulectomy, or capsulotomy) at any time prior to the study.
3. Has any abnormalities/conditions in the affected shoulder that would be potentially confounding as determined by the central MRI review committee grading criteria.
4. Has a prosthesis or replacement of right or left shoulder, elbow, wrist, and/or hand.
5. Has systemic conditions (malignancy, hypertension, diabetes, thyroid disease, thrombosis, physical impairment, infection, significant medical condition) that restricts study participation.
6. Has any contraindications for MRI (implant containing metal, internal metallic object, permanent cosmetics/make-up/tattoos, claustrophobia, anemia, uncontrolled hypertension, epilepsy, asthma, sickle cell disease) as determined by the technologist, the radiologist, and/or investigator performing the imaging, with exemption of the area to be treated/reviewed.
7. Has a known coagulation disorder or is taking any medications that would increase the risk of bleeding (except <150 milligrams of aspirin daily), 7 days prior to first injection and for the duration of the study.
8. Has received oral or parenteral steroids for any reason within 3 weeks before the Screening Visit.
9. Has, at any time, received collagenase for the treatment of adhesive capsulitis (including participant who received treatment in Study AUX-CC-870 or AUX-CC-871).
10. Has received treatment with an investigational product within 30 days (or 5 half lives, whichever is longer) of the screening visit.
11. Has received collagenase treatments (for example, Santyl® ointment and/or XIAFLEX/XIAPEX®) for any other indication within 30 days prior to study treatment administration, or is planning to be treated with collagenase (other than study treatment) at any time during the study.
12. Has donated blood within 30 days prior to the Screening Visit or has plans to donate blood during the study.
13. Has a corrected QT interval (QTc) of ≥ 450 milliseconds (ms) for male participant or ≥470 ms for female participant on the screening electrocardiogram (ECG).
14. Is from a vulnerable population, as defined by the US Code of Federal Regulations (CFR) Title 45, Part 46, Section 46.111(b) and other local and national regulations, including but not limited to, employees (temporary, part-time, full-time, etc) or a family member of the research staff conducting the study, or of the sponsor, or of the contract research organization, or of the Institutional Review Board (IRB)/Independent Ethics Committee (IEC).
15. Has concurrent diseases that might interfere with the conduct of the study, confound the interpretation of the study results, or endanger the participant's well-being, (for example, evidence of any significant hematological, endocrine, cardiovascular, respiratory, neurological, renal, hepatic, or gastrointestinal disease). If there is a history of such disease but the condition has been stable for more than 5 year(s) and is judged by the investigator not to interfere with the participant's participation in the study, the participant may be included, with the documented approval of the Medical Monitor.
16. Has any other condition(s) that, in the investigator's opinion, might indicate the participant to be unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Ortega, MD, Study Director — Endo Pharmaceuticals
Locations (38):
- United States (38):
  - Endo Clinical Trial Site #38, Birmingham, Alabama
  - Endo Clinical Trial Site #24, Birmingham, Alabama
  - Endo Clinical Trial Site #9, Mobile, Alabama
  - Endo Clinical Trial Site #29, Tucson, Arizona
  - Endo Clinical Trial Site #12, Encinitas, California
  - Endo Clinical Trial Site #16, Huntington Beach, California
  - Endo Clinical Trial Site #18, La Mesa, California
  - Endo Clinical Trial Site #14, Pasadena, California
  - Endo Clinical Trial Site #37, Denver, Colorado
  - Endo Clinical Trial Site #33, Bradenton, Florida
  - Endo Clinical Trial Site #3, Clearwater, Florida
  - Endo Clinical Trial Site #32, Clermont, Florida
  - Endo Clinical Trial Site #13, DeLand, Florida
  - Endo Clinical Trial Site #1, Fort Lauderdale, Florida
  - Endo Clinical Trial Site #2, Tampa, Florida
  - Endo Clinical Trial Site #20, Winter Park, Florida
  - Endo Clinical Trial Site #34, Dalton, Georgia
  - Endo Clinical Trial Site #26, Lawrenceville, Georgia
  - Endo Clinical Trial Site #30, Newnan, Georgia
  - Endo Clinical Trial Site #28, Stockbridge, Georgia
  - Endo Clinical Trial Site #31, Oak Brook, Illinois
  - Endo Clinical Trial Site #35, New Orleans, Louisiana
  - Endo Clinical Trial Site #8, Lincoln, Nebraska
  - Endo Clinical Trial Site #10, Stony Brook, New York
  - Endo Clinical Trial Site #21, Durham, North Carolina
  - Endo Clinical Trial Site #36, Mooresville, North Carolina
  - Endo Clinical Trial Site #6, Dayton, Ohio
  - Endo Clinical Trial Site #11, Altoona, Pennsylvania
  - Endo Clinical Trial Site #7, Indiana, Pennsylvania
  - Endo Clinical Trial Site #5, State College, Pennsylvania
  - Endo Clinical Trial Site #17, Bedford, Texas
  - Endo Clinical Trial Site #19, Bellaire, Texas
  - Endo Clinical Trial Site #15, Fort Worth, Texas
  - Endo Clinical Trial Site #27, Georgetown, Texas
  - Endo Clinical Trial Site #25, Laredo, Texas
  - Endo Clinical Trial Site #23, Plano, Texas
  - Endo Clinical Trial Site #22, Plano, Texas
  - Endo Clinical Trial Site #4, Danville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

RESULTS

PARTICIPANT FLOW:
Groups:
- EN3835: Participants received EN3835 (up to 1.74 mg total) by pericapsular (periarticular) injection in up to 3 treatment sessions at least 21 days apart.
- Placebo: Participants received placebo by pericapsular (periarticular) injection in up to 3 treatment sessions at least 21 days apart.
Period: Overall Study
Arm/Group | EN3835 | Placebo
Started | 102 | 96
Received at Least 1 Dose of Study Drug | 101 | 94
Completed | 84 | 80
Not Completed | 18 | 16
Not completed — Adverse Event | 6 | 2
Not completed — Withdrawal by Subject | 7 | 6
Not completed — Lost to Follow-up | 3 | 5
Not completed — Not Treated | 1 | 2
Not completed — Other Than Specified | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 injection of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | EN3835 | Placebo | Total
Number analyzed (Participants) | 101 | 94 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.76 (7.565) | 55.50 (7.806) | 54.59 (7.712)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 66 | 131
  Male | 36 | 28 | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 4 | 6 | 10
  Black | 12 | 11 | 23
  White | 82 | 72 | 154
  Other Race | 2 | 2 | 4
  Multiple Race | 0 | 1 | 1
  Hispanic or Latino | 14 | 16 | 30
  Not Hispanic or Latino | 87 | 78 | 165

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Adapted American Shoulder and Elbow Surgeons Shoulder Assessment Form (ASES) Composite Score for the Affected Shoulder at Day 95
Description: Adapted ASES is a self-administered participant reported outcome measure, divided into 2 sections: pain and function. Pain subscale is a single item, 11-point numeric rating scale, ranging from 0 (no pain at all) to 10 (worst pain), calculated as 10 - pain raw score and multiplying by 5, score ranging from 0 (worst pain) to 50 (no pain). Function subscale consists of 10 activities, 4-point ordinal scale about their ability to do the activity with the affected arm, ranging from 0 (unable to do) to 3 (not difficult), calculated by multiplying total score for 10 items by 5 and then dividing it by 3, score range of 0 (no function) to 50 (full function).
  Adapted ASES composite score is the sum of the pain subscale score (50% of the composite score) and function subscale score (50% of the composite score), score range of 0 (worst pain) to 100 (least pain). Positive change from Baseline score means an improvement in pain and/or shoulder function.
Time Frame: Baseline, Day 95
Population: Modified intent-to-treat population included all randomized participants who received at least 1 injection of study treatment and who had a valid baseline adapted ASES composite score in the affected shoulder and at least 1 valid adapted ASES composite score after the injection of the study treatment and had both Baseline and Day 95 measurements. Here, overall number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 84 | 82
score on a scale | 41.35 (22.432) | 41.16 (21.942)
Statistical Analysis 1: Comparison: EN3835 vs Placebo; Mixed Model Repeated Measures (MMRM) was performed to estimate the change from Baseline treatment effect of the adapted ASES composite score in the affected shoulder comparing EN3835 to placebo treatment; Test type: Other; p = 0.659, MMRM — Considered significant if p-value is less than 0.05; Least Square Mean Treatment Difference = 1.386, 95% CI 2-sided [-4.804 to 7.577] — The model included treatment, visit and interaction of treatment, visit as fixed effects, Baseline as a covariate, and repeated measures with visit/participant. Treatment difference: EN3835 - Placebo

2. Secondary Outcome: Change From Baseline in Passive Range of Motion (PROM) for Forward Flexion in the Affected Shoulder
Description: PROM for forward flexion was measured using a goniometer. Positive change from Baseline means an improvement.
Time Frame: Baseline, Days 22, 43, 64, and 95
Population: Modified intent-to-treat population included all randomized participants who received at least 1 injection of study treatment and who had a valid baseline adapted ASES composite score in the affected shoulder and at least 1 valid adapted ASES composite score after the injection of the study treatment. Here, number analyzed = participants evaluable at specified time-point (had both Baseline and measurements at specified timepoints).
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 91 | 86
degrees
  Day 22 | 19.1 (24.88) | 13.9 (22.40)
  Day 43: number analyzed (Participants) | 86 | 82
  Day 43 | 25.6 (26.89) | 21.4 (20.14)
  Day 64: number analyzed (Participants) | 85 | 79
  Day 64 | 31.4 (26.31) | 27.3 (23.68)
  Day 95: number analyzed (Participants) | 84 | 83
  Day 95 | 32.8 (25.59) | 29.7 (27.08)

3. Secondary Outcome: Change From Baseline in PROM for Internal Rotation in the Affected Shoulder
Description: PROM for internal rotation was measured using a goniometer and a spinal level. Positive change from Baseline means an improvement.
Time Frame: Baseline, Days 22, 43, 64, and 95
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 90 | 83
degrees
  Day 22 | 6.9 (23.95) | 7.0 (17.94)
  Day 43: number analyzed (Participants) | 85 | 80
  Day 43 | 11.0 (25.97) | 12.4 (19.92)
  Day 64: number analyzed (Participants) | 84 | 76
  Day 64 | 18.0 (24.65) | 18.3 (21.95)
  Day 95: number analyzed (Participants) | 83 | 80
  Day 95 | 19.9 (22.59) | 21.6 (23.11)

4. Secondary Outcome: Change From Baseline in PROM for External Rotation in the Affected Shoulder
Description: PROM for external rotation was measured using a goniometer. Positive change from Baseline means an improvement.
Time Frame: Baseline, Days 22, 43, 64, and 95
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 91 | 86
degrees
  Day 22 | 7.3 (19.39) | 8.8 (15.61)
  Day 43: number analyzed (Participants) | 86 | 82
  Day 43 | 11.2 (20.98) | 14.5 (18.87)
  Day 64: number analyzed (Participants) | 85 | 79
  Day 64 | 17.4 (24.87) | 17.8 (17.87)
  Day 95: number analyzed (Participants) | 84 | 83
  Day 95 | 19.1 (21.24) | 19.2 (18.20)

5. Secondary Outcome: Change From Baseline in PROM for Abduction in the Affected Shoulder
Description: PROM for abduction was measured using a goniometer. Positive change from Baseline means an improvement.
Time Frame: Baseline, Days 22, 43, 64, and 95
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 90 | 86
degrees
  Day 22 | 15.6 (28.47) | 13.1 (23.89)
  Day 43: number analyzed (Participants) | 86 | 82
  Day 43 | 29.6 (30.19) | 18.9 (27.13)
  Day 64: number analyzed (Participants) | 85 | 79
  Day 64 | 35.6 (36.76) | 31.1 (29.27)
  Day 95: number analyzed (Participants) | 84 | 83
  Day 95 | 42.1 (38.17) | 36.0 (33.35)

6. Secondary Outcome: Change From Baseline in PROM for Shoulder Extension in the Affected Shoulder
Description: PROM for shoulder extension was measured using a goniometer. Positive change from Baseline means an improvement.
Time Frame: Baseline, Days 22, 43, 64, and 95
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 91 | 86
degrees
  Day 22 | 3.9 (16.51) | 5.7 (13.54)
  Day 43: number analyzed (Participants) | 86 | 82
  Day 43 | 8.0 (18.34) | 9.2 (16.93)
  Day 64: number analyzed (Participants) | 85 | 79
  Day 64 | 15.2 (18.44) | 12.0 (17.23)
  Day 95: number analyzed (Participants) | 84 | 83
  Day 95 | 20.3 (18.30) | 14.7 (17.15)

7. Secondary Outcome: Change From Baseline in PROM for Forward Flexion in the Affected Shoulder Compared to the Contralateral (Unaffected) Shoulder at Baseline
Description: PROM for forward flexion was measured using a goniometer. PROM measurements for the contralateral (unaffected) shoulder were taken at Baseline. PROM measurements of the affected shoulder were take at Baseline, Days 22, 43, 64, and 95.
  Baseline Value = Measurement at Baseline in Affected Shoulder- Measurement at Baseline Contralateral Unaffected Shoulder
  Change from baseline was calculated as:
  (Measurement at Visit in Affected Shoulder - Measurement at Baseline Contralateral Shoulder) - Baseline Value
Time Frame: Baseline, Days 22, 43, 64, and 95
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 91 | 86
degrees
  Day 22 | -34.48 (29.067) | -37.33 (27.179)
  Day 43: number analyzed (Participants) | 86 | 82
  Day 43 | -28.34 (27.939) | -30.24 (26.369)
  Day 64: number analyzed (Participants) | 85 | 79
  Day 64 | -22.14 (27.983) | -23.01 (24.200)
  Day 95: number analyzed (Participants) | 84 | 83
  Day 95 | -20.82 (26.245) | -21.06 (25.198)

8. Secondary Outcome: Change From Baseline in PROM for Internal Rotation in the Affected Shoulder Compared to the Contralateral (Unaffected) Shoulder at Baseline
Description: PROM for internal rotation was measured using a goniometer and a spinal level. PROM measurements for the contralateral (unaffected) shoulder were taken at Baseline. PROM measurements of the affected shoulder were take at Baseline, Days 22, 43, 64, and 95.
  Baseline Value = Measurement at Baseline in Affected Shoulder- Measurement at Baseline Contralateral Unaffected Shoulder
  Change from baseline was calculated as:
  (Measurement at Visit in Affected Shoulder - Measurement at Baseline Contralateral Shoulder) - Baseline Value
Time Frame: Baseline, Days 22, 43, 64, and 95
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 90 | 83
degrees
  Day 22 | -30.76 (24.692) | -28.51 (24.930)
  Day 43: number analyzed (Participants) | 85 | 80
  Day 43 | -26.81 (24.950) | -22.03 (24.311)
  Day 64: number analyzed (Participants) | 84 | 76
  Day 64 | -20.50 (21.561) | -16.88 (24.096)
  Day 95: number analyzed (Participants) | 83 | 80
  Day 95 | -18.22 (21.444) | -13.49 (26.037)

9. Secondary Outcome: Change From Baseline in PROM for External Rotation in the Affected Shoulder Compared to the Contralateral (Unaffected) Shoulder at Baseline
Description: PROM for external rotation was measured using a goniometer PROM measurements for the contralateral (unaffected) shoulder were taken at Baseline. PROM measurements of the affected shoulder were take at Baseline, Days 22, 43, 64, and 95.
  Baseline Value = Measurement at Baseline in Affected Shoulder- Measurement at Baseline Contralateral Unaffected Shoulder
  Change from baseline was calculated as:
  (Measurement at Visit in Affected Shoulder - Measurement at Baseline Contralateral Shoulder) - Baseline Value
Time Frame: Baseline, Days 22, 43, 64, and 95
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 91 | 86
degrees
  Day 22 | -35.12 (22.928) | -35.49 (23.027)
  Day 43: number analyzed (Participants) | 86 | 82
  Day 43 | -31.30 (25.102) | -29.40 (25.727)
  Day 64: number analyzed (Participants) | 85 | 79
  Day 64 | -24.46 (26.063) | -26.08 (24.494)
  Day 95: number analyzed (Participants) | 84 | 83
  Day 95 | -22.94 (22.153) | -25.06 (23.844)

10. Secondary Outcome: Change From Baseline in PROM for Abduction in the Affected Shoulder Compared to the Contralateral (Unaffected) Shoulder at Baseline
Description: PROM for abduction was measured using a goniometer. PROM measurements for the contralateral (unaffected) shoulder were taken at Baseline. PROM measurements of the affected shoulder were take at Baseline, Days 22, 43, 64, and 95.
  Baseline Value = Measurement at Baseline in Affected Shoulder- Measurement at Baseline Contralateral Unaffected Shoulder
  Change from baseline was calculated as:
  (Measurement at Visit in Affected Shoulder - Measurement at Baseline Contralateral Shoulder) - Baseline Value
Time Frame: Baseline, Days 22, 43, 64, and 95
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 90 | 86
degrees
  Day 22 | -54.90 (40.162) | -57.56 (35.565)
  Day 43: number analyzed (Participants) | 86 | 82
  Day 43 | -41.37 (39.918) | -53.17 (36.106)
  Day 64: number analyzed (Participants) | 85 | 79
  Day 64 | -34.87 (39.860) | -41.48 (37.136)
  Day 95: number analyzed (Participants) | 84 | 83
  Day 95 | -28.91 (41.483) | -36.54 (41.288)

11. Secondary Outcome: Change From Baseline in PROM for Shoulder Extension in the Affected Shoulder Compared to the Contralateral (Unaffected) Shoulder at Baseline
Description: PROM for shoulder extension was measured using a goniometer. PROM measurements for the contralateral (unaffected) shoulder were taken at Baseline. PROM measurements of the affected shoulder were take at Baseline, Days 22, 43, 64, and 95.
  Baseline Value = Measurement at Baseline in Affected Shoulder- Measurement at Baseline Contralateral Unaffected Shoulder
  Change from baseline was calculated as:
  (Measurement at Visit in Affected Shoulder - Measurement at Baseline Contralateral Shoulder) - Baseline Value
Time Frame: Baseline, Days 22, 43, 64, and 95
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 91 | 86
degrees
  Day 22 | -18.82 (21.558) | -17.11 (19.106)
  Day 43: number analyzed (Participants) | 86 | 82
  Day 43 | -14.99 (22.313) | -14.01 (20.363)
  Day 64: number analyzed (Participants) | 85 | 79
  Day 64 | -7.97 (22.633) | -9.91 (18.869)
  Day 95: number analyzed (Participants) | 84 | 83
  Day 95 | -2.87 (20.756) | -7.33 (17.676)

12. Secondary Outcome: Change From Baseline in Active Range of Motion (AROM) for Forward Flexion in the Affected Shoulder
Description: AROM for forward flexion was measured using a goniometer. Positive change from Baseline means an improvement.
Time Frame: Baseline, Days 22, 43, 64, and 95
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 91 | 86
degrees
  Day 22 | 13.6 (26.28) | 13.0 (26.55)
  Day 43: number analyzed (Participants) | 86 | 82
  Day 43 | 21.9 (30.00) | 22.3 (26.17)
  Day 64: number analyzed (Participants) | 85 | 79
  Day 64 | 27.7 (25.47) | 29.6 (28.85)
  Day 95: number analyzed (Participants) | 84 | 83
  Day 95 | 31.7 (25.31) | 30.1 (31.20)

13. Secondary Outcome: Change From Baseline in AROM for Internal Rotation in the Affected Shoulder
Description: AROM for internal rotation was measured using a goniometer and a spinal level. Positive change from Baseline means an improvement.
Time Frame: Baseline, Days 22, 43, 64, and 95
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 90 | 83
degrees
  Day 22 | 7.5 (20.45) | 5.8 (19.12)
  Day 43: number analyzed (Participants) | 85 | 80
  Day 43 | 9.1 (22.13) | 10.2 (20.40)
  Day 64: number analyzed (Participants) | 84 | 76
  Day 64 | 18.4 (22.44) | 17.5 (21.55)
  Day 95: number analyzed (Participants) | 83 | 80
  Day 95 | 19.6 (21.99) | 21.6 (23.87)

14. Secondary Outcome: Change From Baseline in AROM for External Rotation in the Affected Shoulder
Description: AROM for external rotation was measured using a goniometer. Positive change from Baseline means an improvement.
Time Frame: Baseline, Days 22, 43, 64, and 95
Population: All randomized participants who received at least 1 injection of study treatment who had a valid baseline adapted ASES composite score in the affected shoulder and at least 1 valid adapted ASES composite score after the injection of the study treatment and had both Baseline and measurements at specified timepoints.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 91 | 85
degrees
  Day 22 | 5.3 (16.85) | 5.6 (14.79)
  Day 43: number analyzed (Participants) | 86 | 82
  Day 43 | 8.7 (19.59) | 10.0 (19.12)
  Day 64: number analyzed (Participants) | 85 | 79
  Day 64 | 13.9 (22.18) | 15.4 (21.65)
  Day 95: number analyzed (Participants) | 84 | 83
  Day 95 | 16.8 (21.67) | 16.1 (21.00)

15. Secondary Outcome: Change From Baseline in AROM for Abduction in the Affected Shoulder
Description: AROM for abduction was measured using a goniometer. Positive change from Baseline means an improvement.
Time Frame: Baseline, Days 22, 43, 64, and 95
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 91 | 85
degrees
  Day 22 | 14.2 (30.75) | 13.7 (23.17)
  Day 43: number analyzed (Participants) | 86 | 82
  Day 43 | 26.6 (37.79) | 22.2 (27.93)
  Day 64: number analyzed (Participants) | 85 | 79
  Day 64 | 37.2 (35.60) | 33.3 (30.53)
  Day 95: number analyzed (Participants) | 84 | 83
  Day 95 | 42.0 (37.71) | 39.8 (31.79)

16. Secondary Outcome: Change From Baseline in AROM for Shoulder Extension in the Affected Shoulder
Description: AROM for shoulder extension was measured using a goniometer. Positive change from Baseline means an improvement.
Time Frame: Baseline, Days 22, 43, 64, and 95
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 91 | 83
degrees
  Day 22 | 7.0 (17.37) | 8.5 (15.84)
  Day 43: number analyzed (Participants) | 86 | 81
  Day 43 | 13.7 (21.63) | 12.0 (16.72)
  Day 64: number analyzed (Participants) | 85 | 77
  Day 64 | 16.2 (19.29) | 15.3 (16.70)
  Day 95: number analyzed (Participants) | 84 | 82
  Day 95 | 19.7 (19.91) | 17.3 (17.17)

17. Secondary Outcome: Change From Baseline in AROM for Forward Flexion in the Affected Shoulder Compared to the Contralateral (Unaffected) Shoulder at Baseline
Description: AROM for forward flexion was measured using a goniometer. AROM measurements for the contralateral (unaffected) shoulder were taken at Baseline. AROM measurements of the affected shoulder were take at Baseline, Days 22, 43, 64, and 95.
  Baseline Value = Measurement at Baseline in Affected Shoulder- Measurement at Baseline Contralateral Unaffected Shoulder
  Change from baseline was calculated as:
  (Measurement at Visit in Affected Shoulder - Measurement at Baseline Contralateral Shoulder) - Baseline Value
Time Frame: Baseline, Days 22, 43, 64, and 95
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 91 | 86
degrees
  Day 22 | -38.34 (30.007) | -40.72 (24.602)
  Day 43: number analyzed (Participants) | 86 | 82
  Day 43 | -31.00 (29.397) | -32.17 (24.879)
  Day 64: number analyzed (Participants) | 85 | 79
  Day 64 | -23.62 (29.115) | -23.82 (23.083)
  Day 95: number analyzed (Participants) | 84 | 83
  Day 95 | -19.83 (26.729) | -23.39 (24.774)

18. Secondary Outcome: Change From Baseline in AROM for Internal Rotation in the Affected Shoulder Compared to the Contralateral (Unaffected) Shoulder at Baseline
Description: AROM for internal rotation was measured using a goniometer and a spinal level. AROM measurements for the contralateral (unaffected) shoulder were taken at Baseline. AROM measurements of the affected shoulder were take at Baseline, Days 22, 43, 64, and 95.
  Baseline Value = Measurement at Baseline in Affected Shoulder- Measurement at Baseline Contralateral Unaffected Shoulder
  Change from baseline was calculated as:
  (Measurement at Visit in Affected Shoulder - Measurement at Baseline Contralateral Shoulder) - Baseline Value
Time Frame: Baseline, Days 22, 43, 64, and 95
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 90 | 86
degrees
  Day 22 | -30.53 (24.699) | -27.94 (24.757)
  Day 43: number analyzed (Participants) | 86 | 82
  Day 43 | -29.78 (24.728) | -23.45 (24.923)
  Day 64: number analyzed (Participants) | 85 | 79
  Day 64 | -20.57 (23.335) | -16.99 (24.708)
  Day 95: number analyzed (Participants) | 84 | 83
  Day 95 | -19.27 (23.646) | -12.66 (27.685)

19. Secondary Outcome: Change From Baseline in AROM for External Rotation in the Affected Shoulder Compared to the Contralateral (Unaffected) Shoulder at Baseline
Description: AROM for external rotation was measured using a goniometer. AROM measurements for the contralateral (unaffected) shoulder were taken at Baseline. AROM measurements of the affected shoulder were take at Baseline, Days 22, 43, 64, and 95.
  Baseline Value = Measurement at Baseline in Affected Shoulder- Measurement at Baseline Contralateral Unaffected Shoulder
  Change from baseline was calculated as:
  (Measurement at Visit in Affected Shoulder - Measurement at Baseline Contralateral Shoulder) - Baseline Value
Time Frame: Baseline, Days 22, 43, 64, and 95
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 91 | 85
degrees
  Day 22 | -34.78 (25.743) | -35.82 (22.666)
  Day 43: number analyzed (Participants) | 86 | 82
  Day 43 | -31.07 (29.543) | -31.23 (23.379)
  Day 64: number analyzed (Participants) | 85 | 79
  Day 64 | -25.31 (28.454) | -25.84 (26.291)
  Day 95: number analyzed (Participants) | 84 | 83
  Day 95 | -22.52 (26.313) | -25.42 (26.075)

20. Secondary Outcome: Change From Baseline in AROM for Abduction in the Affected Shoulder Compared to the Contralateral (Unaffected) Shoulder at Baseline
Description: AROM for abduction was measured using a goniometer. AROM measurements for the contralateral (unaffected) shoulder were taken at Baseline. AROM measurements of the affected shoulder were take at Baseline, Days 22, 43, 64, and 95.
  Baseline Value = Measurement at Baseline in Affected Shoulder- Measurement at Baseline Contralateral Unaffected Shoulder
  Change from baseline was calculated as:
  (Measurement at Visit in Affected Shoulder - Measurement at Baseline Contralateral Shoulder) - Baseline Value
Time Frame: Baseline, Days 22, 43, 64, and 95
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 91 | 85
degrees
  Day 22 | -58.41 (38.888) | -57.28 (36.353)
  Day 43: number analyzed (Participants) | 86 | 82
  Day 43 | -46.14 (41.198) | -49.32 (34.988)
  Day 64: number analyzed (Participants) | 85 | 79
  Day 64 | -35.08 (36.868) | -39.82 (38.397)
  Day 95: number analyzed (Participants) | 84 | 83
  Day 95 | -30.74 (38.227) | -33.01 (39.718)

21. Secondary Outcome: Change From Baseline in AROM for Shoulder Extension in the Affected Shoulder Compared to the Contralateral (Unaffected) Shoulder at Baseline
Description: AROM for shoulder extension was measured using a goniometer. AROM measurements for the contralateral (unaffected) shoulder were taken at Baseline. AROM measurements of the affected shoulder were take at Baseline, Days 22, 43, 64, and 95.
  Baseline Value = Measurement at Baseline in Affected Shoulder- Measurement at Baseline Contralateral Unaffected Shoulder
  Change from baseline was calculated as:
  (Measurement at Visit in Affected Shoulder - Measurement at Baseline Contralateral Shoulder) - Baseline Value
Time Frame: Baseline, Days 22, 43, 64, and 95
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 91 | 84
degrees
  Day 22 | -13.65 (19.893) | -15.25 (21.385)
  Day 43: number analyzed (Participants) | 86 | 82
  Day 43 | -7.55 (20.771) | -11.65 (20.674)
  Day 64: number analyzed (Participants) | 85 | 78
  Day 64 | -4.29 (20.214) | -6.94 (20.775)
  Day 95: number analyzed (Participants) | 84 | 83
  Day 95 | -1.00 (18.904) | -5.34 (20.922)

22. Secondary Outcome: Change From Baseline in the Adapted ASES Composite Score
Description: The adapted ASES is a self-administered participant reported outcome measure, divided into 2 sections: pain and function. Pain subscale is a single item, 11-point numeric rating scale, ranging from (no pain at all) to 10 (worst pain), calculated as 10 - pain raw score and multiplying by 5, score ranging from 0 (worst pain) to 50 (no pain). Function subscale consists of 10 activities, 4-point ordinal scale about their ability to do the activity with the affected arm, ranging from 0 (unable to do) to 3 (not difficult), calculated by multiplying the total score for 10 items by 5 and then dividing it by 3, score ranging from 0 (no function) to 50 (full function).
  The adapted ASES composite score is the sum of the pain subscale score (50% of the composite score) and function subscale score (50% of the composite score). The range for composite score is 0 (worst pain) to 100 (least pain). Positive change from Baseline score means an improvement in pain and/or shoulder function.
Time Frame: Baseline, Day 22, 43, and 64
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 91 | 85
score on a scale
  Day 22 | 14.87 (15.684) | 15.96 (14.269)
  Day 43: number analyzed (Participants) | 88 | 83
  Day 43 | 25.15 (21.532) | 21.77 (18.199)
  Day 64: number analyzed (Participants) | 83 | 80
  Day 64 | 38.21 (22.837) | 34.98 (21.222)

23. Secondary Outcome: Change From Baseline in the Adapted ASES Function Subscale Score
Description: The adapted ASES function subscale consists of 10 activities, 4-point ordinal scale about their ability to do the activity with the affected arm, ranging from 0 (unable to do) to 3 (not difficult), calculated by multiplying the total score for 10 items by 5 and then dividing it by 3, score ranging from 0 (worst no function) to 50 (full function).
  Positive change from Baseline score means an improvement in shoulder function.
Time Frame: Baseline, Day 22, 43, 64, and 95
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 91 | 85
score on a scale
  Day 22 | 7.56 (8.245) | 7.96 (7.388)
  Day 43: number analyzed (Participants) | 88 | 83
  Day 43 | 12.82 (10.365) | 11.77 (9.964)
  Day 64: number analyzed (Participants) | 83 | 80
  Day 64 | 19.60 (12.127) | 17.98 (11.337)
  Day 95: number analyzed (Participants) | 84 | 82
  Day 95 | 21.05 (11.538) | 20.73 (11.823)

24. Secondary Outcome: Change From Baseline in the Adapted ASES Pain Subscale Score
Description: The adapted ASES pain subscale is a single item, 11-point numeric rating scale, ranging from (no pain at all) to 10 (worst pain), calculated as 10 - pain raw score and multiplying by 5, score ranging from 0 (worst pain) to 50 (no pain). Positive change from Baseline score means an improvement in shoulder pain.
Time Frame: Baseline, Day 22, 43, 64, and 95
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 91 | 85
score on a scale
  Day 22 | 7.3 (9.61) | 8.0 (9.49)
  Day 43: number analyzed (Participants) | 88 | 83
  Day 43 | 12.3 (12.73) | 10.0 (11.87)
  Day 64: number analyzed (Participants) | 83 | 80
  Day 64 | 18.6 (12.67) | 17.0 (12.29)
  Day 95: number analyzed (Participants) | 84 | 82
  Day 95 | 20.3 (13.11) | 20.4 (12.28)

25. Secondary Outcome: Change From Baseline in the Pain Upon Movement (PUM) Scale Score for the Affected Shoulder
Description: The PUM scale is a single item 11-point numerical rating scale of pain in the affected shoulder after AROM forward flexion, internal rotation, external rotation, abduction, and shoulder extension on a scale from 0 (no pain at all) to 10 (pain as bad as it can be). A decrease from Baseline indicates improvement.
Time Frame: Baseline, Days 64 and 95
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 88 | 82
score on a scale
  Day 64: number analyzed (Participants) | 88 | 77
  Day 64 | -3.6 (2.60) | -3.0 (2.72)
  Day 95: number analyzed (Participants) | 84 | 82
  Day 95 | -4.1 (2.59) | -3.8 (2.96)

26. Secondary Outcome: Change From Baseline in Patient-reported Global Severity of Adhesive Capsulitis Scale
Description: The Patient-reported Global Severity of Adhesive Capsulitis is a single item, 11-point numerical rating scale that asks participants to rate the overall severity of their adhesive capsulitis symptoms on a scale from 0 (no severity) to 10 (severe as can be). A decrease from Baseline indicates improvement.
Time Frame: Baseline, Day 22, 43, 64, and 95
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 90 | 84
score on a scale
  Day 22 | -1.8 (1.84) | -1.5 (1.87)
  Day 43: number analyzed (Participants) | 85 | 83
  Day 43 | -3.0 (2.21) | -2.3 (2.16)
  Day 64: number analyzed (Participants) | 84 | 80
  Day 64 | -4.0 (2.41) | -3.6 (2.61)
  Day 95: number analyzed (Participants) | 84 | 82
  Day 95 | -4.4 (2.48) | -4.0 (2.87)

27. Secondary Outcome: Patient-reported Change in Severity of Adhesive Capsulitis Scale
Description: The Patient-reported Change in Severity of Adhesive Capsulitis is a questionnaire that asks participants if their adhesive capsulitis symptoms are "Better, About the Same, or Worse" since the last time the questionnaire was administered. Participants who reported that their symptoms are better or worse are then asked to rate the change in their symptoms on a 7-point ordinal scale for worse and better severity. An overall severity of worse was rated from 0 (almost the same, hardly worse at all) to -6 (a very great deal worse). An overall severity of better was rated from 0 (almost the same, hardly better at all) to 6 (a very great deal better).
  Only participants with a response of 'Worse' or 'Better' were analyzed. Participants with an overall severity response of 'About the same' were excluded from the summary table below. For overall worse severity, a lower score indicated a worse outcome. For overall better severity, a higher score indicated a better outcome.
Time Frame: Days 22, 43, 64 and 95
Population: Modified intent-to-treat population included all randomized participants who received at least 1 injection of study treatment and who had a valid baseline adapted ASES composite score in the affected shoulder and at least 1 valid adapted ASES composite score after the injection of the study treatment. Here, number analyzed = participants evaluable at specified time-point (had measurement at specified timepoint).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 72 | 69
score on a scale
  Day 22: Worse Severity: number analyzed (Participants) | 5 | 6
  Day 22: Worse Severity | -3.4 (1.52) | -3.2 (2.23)
  Day 22: Better Severity: number analyzed (Participants) | 57 | 51
  Day 22: Better Severity | 2.4 (1.40) | 2.5 (1.29)
  Day 43: Worse Severity: number analyzed (Participants) | 3 | 4
  Day 43: Worse Severity | -3.3 (1.53) | -4.0 (2.16)
  Day 43: Better Severity: number analyzed (Participants) | 65 | 56
  Day 43: Better Severity | 3.4 (1.46) | 3.6 (1.44)
  Day 64: Worse Severity: number analyzed (Participants) | 0 | 4
  Day 64: Worse Severity |  | -4.8 (0.50)
  Day 64: Better Severity: number analyzed (Participants) | 69 | 64
  Day 64: Better Severity | 4.5 (1.29) | 4.2 (1.40)
  Day 95: Worse Severity: number analyzed (Participants) | 0 | 4
  Day 95: Worse Severity |  | -3.5 (1.91)
  Day 95: Better Severity: number analyzed (Participants) | 72 | 65
  Day 95: Better Severity | 4.7 (1.27) | 4.7 (1.09)

28. Secondary Outcome: Number of Responders Assessed With Investigator Assessment of Improvement
Description: Investigator assessment of improvement with treatment in the severity of the participant's treated shoulder using a 7-point Likert scale from very much worse (-3) to very much improved (3). A responder was defined as a response of "very much improved", "much improved" or "minimally improved" in the investigator assessment of improvement with treatment.
Time Frame: Days 64 and 95
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 82 | 73
Participants
  Day 64: number analyzed (Participants) | 78 | 69
  Day 64 | 71 | 59
  Day 95 | 80 | 65

29. Secondary Outcome: Number of Responders Assessed by the Subject Satisfaction With Treatment Assessment
Description: Participants rated their satisfaction with treatment on a 7-point Likert scale from very dissatisfied (-3) to very satisfied (3) at specified times for relief of pain in treated shoulder, relief of stiffness in treated shoulder, relief of pain in treated shoulder compared to better shoulder, and relief of stiffness in treated shoulder compared to better shoulder. A responder was defined as a participant with a response of "very satisfied", "satisfied" or "somewhat satisfied" in the satisfaction with treatment.
Time Frame: Days 64 and 95
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 88 | 82
Participants
  Day 64: Pain relief in treated shoulder: number analyzed (Participants) | 88 | 76
  Day 64: Pain relief in treated shoulder | 80 | 60
  Day 64: Stiffness relief in treated shoulder: number analyzed (Participants) | 88 | 76
  Day 64: Stiffness relief in treated shoulder | 74 | 59
  Day 64: Pain relief in treated shoulder compared to better shoulder: number analyzed (Participants) | 88 | 76
  Day 64: Pain relief in treated shoulder compared to better shoulder | 74 | 57
  Day 64: Stiffness relief in treated shoulder compared to better shoulder: number analyzed (Participants) | 88 | 76
  Day 64: Stiffness relief in treated shoulder compared to better shoulder | 73 | 54
  Day 95: Pain relief in treated shoulder: number analyzed (Participants) | 84 | 82
  Day 95: Pain relief in treated shoulder | 73 | 69
  Day 95: Stiffness relief in treated shoulder: number analyzed (Participants) | 84 | 82
  Day 95: Stiffness relief in treated shoulder | 71 | 69
  Day 95: Pain relief in treated shoulder compared to better shoulder: number analyzed (Participants) | 84 | 82
  Day 95: Pain relief in treated shoulder compared to better shoulder | 71 | 68
  Day 95: Stiffness relief in treated shoulder compared to better shoulder: number analyzed (Participants) | 84 | 82
  Day 95: Stiffness relief in treated shoulder compared to better shoulder | 68 | 65

30. Secondary Outcome: Number of Participants Positive for Anti-AUX-I and Anti-AUX-II Antibodies
Description: Serum samples were collected and tested for the presence of anti-AUX-I and anti-AUX-II antibodies.
Time Frame: Day 95
Population: Safety population included all participants who received at least 1 dose of study drug and had an assessment at the specified timepoint. Here, overall number of participants analyzed = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 83 | 72
Participants
  Anti-AUX-I Antibodies | 83 | 3
  Anti-AUX-II Antibodies | 81 | 3

31. Secondary Outcome: Number of Participants Positive for Neutralizing Antibodies
Description: Serum samples were collected and tested for the presence of anti-AUX-I and anti-AUX-II antibodies. Only samples positive for anti-AUX-I and anti-AUX-II antibodies were analyzed for neutralizing antibodies.
Time Frame: Day 95
Population: All participants who received at least 1 dose of study drug, were positive for anti-AUX-I and anti-AUX-II antibodies and had an assessment at the specified timepoint. Here, overall number of participants analyzed = participants evaluable for this outcome measure. Only samples positive for anti-AUX-I and anti-AUX-II antibodies were analyzed for neutralizing antibodies.
Measure: Count of Participants; unit: Participants
Arm/Group | EN3835 | Placebo
Number analyzed (Participants) | 83 | 3
Participants
  Neutralizing AUX-I Antibodies | 31 | 0
  Neutralizing AUX-II Antibodies: number analyzed (Participants) | 81 | 3
  Neutralizing AUX-II Antibodies | 4 | 0

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) through Day 95
Description: Safety population included all participants who received at least 1 dose of study treatment.
Arm/Group | EN3835 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/94
Serious Adverse Events (participants affected / at risk) | 1/101 | 1/94
Other Adverse Events (participants affected / at risk) | 69/101 | 22/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EN3835 (N=101) | Placebo (N=94)
Depression (Psychiatric disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EN3835 (N=101) | Placebo (N=94)
Injection site bruising (General disorders) | 47 | 4
Injection site pain (General disorders) | 23 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 12
Injection site swelling (General disorders) | 14 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT04496167/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/67/NCT04496167/SAP_001.pdf